CLINICAL TRIAL: NCT00484354
Title: Reduction of Acute Renal Failure Associated With Cardiovascular Surgery: A Randomized Study Comparing Sodium Bicarbonate to Normal Saline
Brief Title: Use of Bicarbonate to Reduce the Incidence of Acute Renal Failure After Cardiac Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00002409
Record Dates: First submitted 2007-06-06; First posted 2007-06-08 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-09

CONDITIONS: Kidney Failure, Acute; Renal Replacement Therapy
Keywords: Acute Renal Failure; Cardiac Surgery; Sodium Bicarbonate; Length of Stay; Mortality
MeSH Terms: conditions — Acute Kidney Injury | interventions — Sodium Bicarbonate; Saline Solution; Bicarbonates

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1 (Active Comparator): Bicarbonate administration
  Interventions: Drug: Sodium bicarbonate; Other: Bicarbonate
- 2 (Placebo Comparator): Normal saline administration
  Interventions: Other: Normal saline; Other: Placebo

INTERVENTIONS:
Drug: Sodium bicarbonate — IV bicarbonate given with amount based on patient weight
  Arms: 1
Other: Normal saline — IV Normal saline with volume given determined by patient weight
  Arms: 2
Other: Bicarbonate — IV bicarbonate, dosed by weight
  Arms: 1
Other: Placebo — Normal saline, with volume given based on patient weight
  Arms: 2

SUMMARY:
The purpose of this study is to determine if the incidence of acute renal failure (ARF) in high risk patients who undergo coronary artery bypass grafting (CABG) is reduced by treating patients in the perioperative period with intravenous (IV) sodium bicarbonate. Patients will be randomized in a 50:50 allocation to receive either IV sodium bicarbonate or IV normal saline. The volume of fluid given in each arm of the study is equal. All other interventions in those patients will be according to standard cardiothoracic anesthesia protocol at our institution.

DETAILED DESCRIPTION:
This is a randomized, controlled, single center study in patients felt to be at high risk for ARF following CABG surgery. Patients who have met the selection criteria noted below will be randomized to one of two treatment arms:

I) Patients allocated to the sodium bicarbonate (NaHCO3) arm will receive a 0.150 M NaHCO3 solution prepared in a sterile water base. An initial bolus of 0.150 M NaHCO3 at 5.0 ml/kg will be given over fifteen minutes prior to surgery. Following the bolus, the 0.150 M NaHCO3 infusion will be run at 1.0 ml/kg/hr during the procedure and for six (6) hours afterwards. The NaHCO3 infusion will then be decreased to 0.4 ml/kg/hr for a further twelve (12) hours. The goal in the NaHCO3 arm is to provide a total dose of approximately 2.5-3.0 mEq/kg of sodium bicarbonate. This dose was determined from prior studies and found to lead to a slight increase in the serum bicarbonate level post-operatively. Anecdotally, the metabolic stress of CABG surgery often leads to a decline in the serum bicarbonate level in patients not treated with alkali therapy.

II) Patients allocated to the normal saline (NS) arm will receive an initial bolus consisting of 0.154 M NaCl (NS) at 5.0 ml/kg given over fifteen minutes prior to surgery. Following the bolus, these patients will receive NS (0.154 M) at a rate of 1.0 ml/kg/hour during the procedure and for six (6) hours afterwards. The rate will then be decreased to 0.4 ml/kg/hour for a further twelve (12) hours as done in the NaHCO3 treatment arm above. There will be a maximum rate of infusion of 125 mL/min used in both study arms to avoid volume overload issues in morbidly obese patients.

There will be no other deviation from standard protocol when treating these patients undergoing CABG at our institution. The standard protocol is dictated by both the cardiothoracic surgeons and anesthesiologists involved with each individual case. The purpose of this study is to compare the incidence of ARF (maximal change in SCr) in high risk patients undergoing CABG when treated with either a NS or NaHCO3 maintenance infusion. This study will test the hypothesis that treatment with NaHCO3 may have a protective effect over NS in preventing AFR following CABG in a high risk population.

ELIGIBILITY:
Inclusion Criteria:

* Calculated GFR ≤ 60 ml/min/m2 (MDRD)

OR

* Any combination of two (2) of the following:
* Age ≥ 70
* Complex surgery (any of the following):

  * CABG/Valve
  * Redo operation
  * Deep hypothermic arrest
* ≥ 2 valves
* History of PVD surgery
* EF < 35%
* Presence of diabetes mellitus
* Prior kidney transplant

Exclusion Criteria:

* Age < 18
* Pre-existing ESRD (dialysis patients)
* Pre-op GFR ≤ 15 ml/min/m2
* Pre-op bicarbonate level ≥ 30 mEq/L
* Emergency surgery (unable to effectively consent)
* Pregnancy
* Heart transplant (OHT)
* Aortic surgery (proximal or distal)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2006-05; Primary Completion 2011-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael V. Rocco, MD, Principal Investigator — Wake Forest University School of Medicine, Dept of Internal Medicine, Division of Nephrology
Locations (1):
- Wake Forest University School of Medicine, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- IV Sodium Bicarbonate: IV sodium bicarbonate given with amount based on patient weight
- IV Normal Saline: IV Normal saline with volume given determined by patient weight
Period: Overall Study
Arm/Group | IV Sodium Bicarbonate | IV Normal Saline
Started | 64 | 59
Completed | 63 | 57
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Sodium Bicarbonate | IV Normal Saline | Total
Number analyzed (Participants) | 64 | 59 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.2 (12.6) | 69.7 (13.5) | 70 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 16 | 46
  Male | 34 | 43 | 77
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 9 | 14
  White | 57 | 47 | 104
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 64 | 59 | 123

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Developed Acute Kidney Injury Within 72 Hours
Description: Number (percentage) of patients who developed acute kidney injury within 72 hours, defined by an increase in serum creatinine level of 0.3 mg/dl from baseline
Time Frame: 72 hours post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | IV Sodium Bicarbonate | IV Normal Saline
Number analyzed (Participants) | 63 | 57
Participants | 17 | 14

2. Secondary Outcome: Change in GFR Over 72 Hours Post Operatively
Description: 25% or greater change in serum creatinine level
Time Frame: 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | IV Sodium Bicarbonate | IV Normal Saline
Number analyzed (Participants) | 63 | 57
Participants | 21 | 21

3. Secondary Outcome: Length of Hospital Stay
Description: Length of hospital stay in days
Time Frame: Until hospital discharge, up to 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IV Sodium Bicarbonate | IV Normal Saline
Number analyzed (Participants) | 63 | 57
days | 14.2 (15.4) | 14.6 (14.4)

4. Secondary Outcome: Number of Participants With Need for Dialysis
Description: Number of participants needing dialysis
Time Frame: Until hospital discharge, up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | IV Sodium Bicarbonate | IV Normal Saline
Number analyzed (Participants) | 63 | 57
Participants | 4 | 5

5. Secondary Outcome: Mortality
Description: Number of patients who died during the hospitalization
Time Frame: Until hospital discharge, up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | IV Sodium Bicarbonate | IV Normal Saline
Number analyzed (Participants) | 63 | 57
Participants | 9 | 10

ADVERSE EVENTS:
Time Frame: Until hospital discharge, up to 30 days
Arm/Group | IV Sodium Bicarbonate | IV Normal Saline
All-Cause Mortality (participants affected / at risk) | 9/63 | 10/57
Serious Adverse Events (participants affected / at risk) | 9/63 | 10/57
Other Adverse Events (participants affected / at risk) | 4/63 | 5/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Sodium Bicarbonate (N=63) | IV Normal Saline (N=57)
Mortality (General disorders) | 9 (9) | 10 (10) — Mortality
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Sodium Bicarbonate (N=63) | IV Normal Saline (N=57)
Dialysis (Renal and urinary disorders) | 4 (4) | 5 (5) — Need for dialysis for treatment of acute kidney injury

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No